CLINICAL TRIAL: NCT01135043
Title: The Impact of the Simple Verbal Intervention for Adequately Collecting Sputum and the Acceptable Specimen Based on Gram Stain, on the Results of Sputum Acid-fast Bacilli Smear Testing
Brief Title: Simple Verbal Intervention for Adequately Collecting Sputum
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Chang-Hoon Lee, Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul Metropolitan Government, Seoul National University Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: acceptable_sputa
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Suspicious for Pulmonary Tuberculosis
Keywords: acceptable sputum; AFB culture; pulmonary tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- education (Experimental): educated with the brochure that contains figure of lung/upper respiratory tract and methods of collecting sputum.
  Interventions: Behavioral: education by brochure
- control (Placebo Comparator): patients with control group are educated about methods of collecting sputum by a physician, only in verbal explanation without brochure.
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: education by brochure — educated with the brochure that contains figure of lung/upper respiratory tract and methods of collecting sputum.
  Arms: education
Behavioral: control — patients with control group are educated about methods of collecting sputum by a physician, only in verbal explanation without brochure
  Arms: control

SUMMARY:
simple verbal intervention with figure of lung and upper respiratory tract will be helpful to adequately collecting sputum.

and in the acceptable specimen based on Gram stain, positivity for AFB stain and culture rate will be higher.

DETAILED DESCRIPTION:
suspicious patients for pulmonary tuberculosis are randomized to control or education group. patients in education group will be educated with the brochure that contains figure of lung/upper respiratory tract and methods of collecting sputum.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* 2009.7~2010.7 patients with suspicious pulmonary tuberculosis who visited Boramae Hospital

Exclusion Criteria:

* on medication for tuberculosis
* patients who medicated with fluoroquinolone within 1month
* patients without consciousness or patients who cannot expectorate sputum
* hemoptysis over 50cc per day
* patients who don't consent on the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
culture result of Mycobacteria in sputum | 8wk after AFB culture

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Lee, MD, Study Chair — Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul Metropolitan Government, Seoul National University Boramae Medical Center
Locations (1):
- Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul Metropolitan Government, Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee YJ, Shin S, Roh EY, Yoon JH, Kim DK, Chung HS, Lee CH. The effectiveness of a brochure describing an acceptable method of sputum collection for tuberculosis testing. Int J Tuberc Lung Dis. 2013 Dec;17(12):1587-9. doi: 10.5588/ijtld.13.0336. PMID 24200273